CLINICAL TRIAL: NCT02323425
Title: Effects of Upper Limb Ischemic Postconditioning on Collateral Circulation in Young Symptomatic Intracranial Atherosclerosis
Brief Title: Effects of Limb Ischemic Postconditioning in Young sICAS
Acronym: EPIC-sICAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Jiaotong University (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Meng Wei, Director, Clinical Research, Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XIANJ-14ZD25
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
Keywords: stroke; Remote ischemic postconditioning; symptomatic atherosclerotic intracranial arterial stenosis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote Ischemic Postconditioning (Experimental): remote ischemic postconditioning（RIPC） treatment was performed by the inflating a cuff around bilateral arms to 180 mmHg with 5 cycles of 3 min inflation and 5 min relax alternation twice a day for the total of 180 consecutive days.
  Interventions: Device: Remote ischemic postconditioning
- Control (No Intervention): Patients in control group will receive foundation treatment. Foundation treatment: including blood vessel expansion、free radical elimination etc during acute phase and aspirin (100-300 mg/d), and atorvastatin (20 mg/d) till the end of the study (180 consecutive days).

INTERVENTIONS:
Device: Remote ischemic postconditioning — Remote ischemic postconditioning（RIPC）treatment was performed by the inflating a cuff around bilateral arms to 180 mmHg with 5 cycles of 3 min inflation and 5 min relax alternation automatically.
  Other Names: limb ischemic postconditioning
  Arms: Remote Ischemic Postconditioning

SUMMARY:
The purpose of this study is to evaluate the protective effects of upper limb ischemic postconditioning on collateral circulationin young symptomatic intracranial atherosclerosis and the baseline characteristics of trial participants, as an open, randomized controlled, prospective controlled trial.

DETAILED DESCRIPTION:
Stroke is a common cardia-cerebrovascular disease with high morbidity, disability and mortality rate. And more and more young patients account for the increasing morbidity. Among them, Symptomatic intracranial atherosclerotic stenosis（sICAS）is a major cause, especially in Asians.

Currently, traditional therapeutic methods present reluctant achievements on reducing stroke recurrence and pose threat on patients'health because of invasive operation and severe side effects. Therefore, other treatment methods are called for urgently. Remote ischemic post-conditioning refers to local or distal ischemia treatment after the occurrence of cerebral ischemia. Prior research has shown that repeatedly ischemic reperfusion have protective effect on lowering the occurrence rate of ischemic events of patients with carotid stenosis. However, in-depth research on cerebral protection and correlation with collateral circulation has not been proven in an open, definitive clinical trial.

Thus, the EPIC-sICAS trial will provide important information on the protective effects of upper limb ischemic post-conditioning on collateral circulation after cerebral Infarction. Hopefully to present us a very meaningful way to improve the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 45 Years old;
2. Symptomatic intracranial atherosclerotic stenosis (sICAS): cranial CTA/MRA/TCD/DSA confirm the diagnosis, patients got ischemic stroke or transient ischemic attack in the brain region supplied by the stenosis artery;
3. National Institutes of Health Stroke Scale(NIHSS) score 0-15
4. Written informed consent was signed.

Exclusion Criteria:

1. Cerebral hemorrhage and other parts of the active bleeding disease;
2. Severe aphasia, unable to express himself;
3. A history of brain tumor, brain trauma, cerebral embolism or other brain lesions;
4. Severe lesions of severe cardiac, liver or kidney disease, malignancy or other systemic organ dysfunction;
5. Blood Pressure< 90 mmHg/60 mmHg or >200 mmHg/110 mmHg after treatment;
6. Dementia and mental illness;
7. Using angiotensin-converting enzyme inhibitors;
8. A history of major surgery or trauma 4 weeks prior to admission;
9. Without informed consent.

Elimination Criteria：

1. Patients with poor compliance，refuse to take regular treatment and examination;
2. patients' condition get exacerbated, with NIHSS score elevate for more than 4.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Mean Change of Collateral Circulation from Baseline and at 6 months | Baseline and at 6 months
  Collateral circulation measured in iconography test: Magnetic Resonance Angiography (MRA)、 Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI)、Arterial spin-labeled (ASL) perfusion magnetic resonance、Transcranial Cerebral Doppler (TCD)、single photon emission computed tomography（SPECT） Baseline was defined as the onset of stroke within 48h. A higher score represents better collateral circulation status functioning.

SECONDARY OUTCOMES:
Mean Change of Symptomatic Recovery | Baseline and at 14 days, 1 month, 6 months, and 1 year
  Functional test: National Institute of Health stroke scale（NIHSS）scores、Activity of Daily Living Scale (ADL) For NIHSS scores, a lower score represents better functioning. For ADL scores, a higher score represents better functioning.
Mean Change of serum vascular endothelial growth factor (VEGF) and basic Fibroblast Growth Factor (bFGF) from Baseline and at 10 days. | Baseline and at 10 days
  A higher amount represents a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: GuoGang Luo, M.D/Ph.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Xunming Ji, M.D/Ph.D, Study Director — Capital Medical University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided